CLINICAL TRIAL: NCT03791450
Title: A Multicenter Big⁃Sample Retrospective Study of Pancreaticoduodenectomy
Brief Title: Investigation of Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaoping, Principal Investigator, Tongji Hospital
Other Study IDs: C201812
Record Dates: First submitted 2018-12-21; First posted 2019-01-02 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pancreaticoduodenectomy: patients underwent pancreaticoduodenectomy in recent ten years.

SUMMARY:
The investigators intend to conduct a multicentre, big-sample, retrospective study to analysis the surgery results of pancreaticoduodenectomy and compare the different suture technique.

DETAILED DESCRIPTION:
For patients with malignant or benign disease of the pancreatic head and periampullary region, pancreaticoduodenectomy is the only potential approach to radical cure. However, pancreaticoduodenectomy is consider as one of the most complex operations associated with a high rate of postoperative complications such as pancreatic fistula, delayed gastric emptying, hemorrhage, abscess, and sepsis. These complications increase the costs associated with pancreaticoduodenectomy. Numerous interventions and techniques have been introduced to decrease the morbidity. But there is little evidence for the superiority of one anastomotic technique over the others. Therefore, investigators intend to conduct a multicentre, big-sample, retrospective study to analysis the surgery results of pancreaticoduodenectomy and compare the different suture technique.

ELIGIBILITY:
Inclusion Criteria:

Patients who had underwent pancreaticoduodenectomy between 2008 to 2018.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had underwent pancreaticoduodenectomy between 2008 to 2018.
Sampling Method: Non-Probability Sample
Enrollment: 10085 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Pancreatic Fistula(POPF) | Within 30 days after surgery
  The frequency of POPF occurs and the POPF will be strictly diagnosis and classified according to IGSPF criteria.

SECONDARY OUTCOMES:
Morbidity | Within 90 days after surgery
  The incidence of operative complications within 90 days after surgery
Mortality | Within 30 days after surgery
  The death occurred within 30 days after surgery
Duration of operation | Intraoperative
  The time of operation count by minute.
Length of hospital stay after surgery | From first day after surgery to release from hospital (anticipate 5 days minimally)
  Days between surgery and hospital discharge
Hospital costs | From first day after surgery to release from hospital (anticipate 5 days minimally)
  The total hospitalization expenses

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China